CLINICAL TRIAL: NCT00482495
Title: A Phase II Trial of Bevacizumab in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Bevacizumab in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Suzanne R. Hayman, M.D., Mayo Clinic
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546757; P30CA015083 (NIH); MC0584 (Other: Mayo Clinic Cancer Center); 05-004261 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bevacizumab; Gene Expression Profiling

INTERVENTIONS:
Biological: bevacizumab
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab may also stop the growth of multiple myeloma by blocking blood flow to the cancer.

PURPOSE: This phase II trial is studying how well bevacizumab works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the hematologic response rate in patients with relapsed or refractory multiple myeloma treated with bevacizumab.
* Determine the proportion of patients who are progression free and have not failed treatment after 1 year.

Secondary

* Determine the toxicity of this drug in these patient.
* Determine the time to disease progression in patients receiving this drug.
* Determine the overall survival and survival at 1 year in patients receiving this drug.

OUTLINE: This is an open-label study.

Patients receive bevacizumab IV on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained for correlative studies at baseline, after course 2, and at 12 weeks. Samples are analyzed for interleukin-6, Flt-1, and VEGF levels.

After completion of study therapy, patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or refractory multiple myeloma
* Measurable or evaluable disease as defined by ≥ 1 of the following:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * Monoclonal protein ≥ 200 mg by 24-hour urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
* No concurrent amyloidosis

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0 or 1

  * ECOG PS 2 based on immobility from myeloma bone disease alone allowed at the discretion of treating physician
* Creatinine ≤ 2.0 mg/dL
* ANC ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Proteinuria ≤ 1 g/dL by 24-hour urine collection (excluding monoclonal protein)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study treatment
* No bleeding diathesis
* No hypertension (defined as BP > 150/100 mm Hg)
* No active bleeding, healing or nonhealing wound, ulcer, or bone fracture (excluding fractures secondary to myeloma)
* No active ulcerative disease including, but not limited to, any of the following:

  * Peptic ulcer disease
  * Ulcerative esophagitis
  * Ulcerative colitis
  * Crohn's disease
* LVEF ≥ 50% by 2-dimensional ECHO or MUGA scan
* No NYHA class III or IV heart disease
* No other active malignancy except for nonmelanoma skin cancer or in situ cervical or breast cancer
* No active infection
* No other comorbidity that would interfere with study compliance
* No transient ischemic attack, cerebrovascular accident, or myocardial infarction within the past year
* No abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within the past 6 months
* No significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 2 prior antimyeloma treatment courses, except for bisphosphonates
* No standard or experimental drug therapy, other than ongoing bisphosphonate treatment and/or epoetin alfa, within the past 28 days
* No experimental non-drug therapy within the past 28 days
* Palliative radiation therapy within the past 28 days allowed provided ≤ 3 sites of bone disease was irradiated
* No prior bevacizumab or other experimental antiangiogenic agents other than thalidomide or lenalidomide
* No minor surgical procedures, fine-needle aspiration, or core biopsies within the past 7 days
* No major surgical procedure or open biopsy within the past 28 days
* No concurrent corticosteroids

  * Chronic steroids ≤ 20 mg/day (prednisone equivalent) for disorders other than myeloma (i.e., adrenal insufficiency, rheumatoid arthritis) allowed
* No other concurrent investigational therapy
* No other concurrent systemic antineoplastic therapy including, but not limited to, the following:

  * Cytotoxic chemotherapy
  * Immunotherapy
  * Hormonal therapy
  * Monoclonal antibody therapy
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Confirmed hematologic response
Progression-free survival at 1 year

SECONDARY OUTCOMES:
Toxicity as measured by NCI CTCAE v3.0
Time to progression
Duration of response
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Hayman, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States